CLINICAL TRIAL: NCT01222689
Title: A Phase 2 Study of AZD6244 Plus Erlotinib for the Second-Line Treatment of Advanced Pancreatic Adenocarcinoma
Brief Title: Selumetinib and Erlotinib Hydrochloride in Treating Patients With Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01266; NCI-2011-01266 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000686634; UCSF-10454; 10454 (Other: UCSF-Mount Zion); 8598 (Other: CTEP); N01CM00070 (NIH); R21CA149939 (NIH)
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride; AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (erlotinib hydrochloride, selumetinib) (Experimental): Patients receive selumetinib PO QD and erlotinib hydrochloride PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Drug: selumetinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given PO
  Other Names: CP-358,774; erlotinib; OSI-774
Drug: selumetinib — Given PO
  Other Names: ARRY-142886; AZD6244
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well giving selumetinib and erlotinib hydrochloride together works in treating patients with locally advanced or metastatic pancreatic cancer that is refractory to chemotherapy. Selumetinib and erlotinib hydrochloride may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

l. To assess overall survival (as measured by median survival and proportion of patients alive at 24 weeks) in patients with advanced pancreatic cancer who have received one prior line of systemic therapy when treated with the combination of AZD6244 (selumetinib) and erlotinib (erlotinib hydrochloride).

SECONDARY OBJECTIVES:

I. Progression-free survival (median progression-free survival [PFS] and proportion of patients with PFS at 12 and 24 weeks).

II. Cancer antigen (CA)19-9 biomarker response (defined as a 50% decline in serum CA19-9 level from baseline in patients with > 2 x upper limit of normal [ULN] CA19-9 measurement).

III. Objective radiographic response by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

IV. Safety and toxicity profile of the combination of AZ6244 and erlotinib.

OUTLINE:

Patients receive selumetinib orally (PO) once daily (QD) and erlotinib hydrochloride PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2-3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven adenocarcinoma of the pancreas
* Patients must have locally advanced unresectable disease not amenable to curative resection or extrapancreatic metastases; patients must have EITHER radiographically measurable disease (defined as at least one lesion that can be accurately measured in at least one dimension [longest diameter to be recorded] as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography [CT] scan) AND/OR a serum CA19-9 measurement > 2 x ULN
* One prior line of systemic therapy for advanced disease (locally advanced or metastatic)

  * The following represent acceptable examples meeting the definition of one prior line of therapy:

    * Gemcitabine as a single agent or in combination with other agents; patients receiving (a) gemcitabine initially alone, with the eventual addition of a second agent; or (b) gemcitabine as part of a combination regimen, followed by gemcitabine alone; are eligible
    * A non-gemcitabine-based regimen, including (but not limited to) leucovorin calcium, fluorouracil, irinotecan hydrochloride, and oxaliplatin (FOLFIRINOX) or any combination of components therein
    * Treatment as part of a clinical trial involving cytotoxic agents, small molecule inhibitors, monoclonal antibodies, and/or immunomodulatory agents
  * For patients with locally advanced disease, prior radiation to the primary tumor is allowable as long as there is clear evidence of disease progression (either radiographic locoregional disease progression and/or a rising CA19-9 level); patients may have received chemotherapy both concurrently and/or sequentially with (either before or after) the radiation and still be eligible for the study, as this would be considered all part of the same course of treatment
  * Treatment given in the adjuvant setting (radiation and/or chemotherapy, given either concurrently or sequentially) does not count as prior therapy as long as progressive disease occurs > 6 months following completion of treatment
* Life expectancy of greater than 8 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Absolute neutrophil count (ANC) >= 1500/uL
* Platelet count >= 100,000/uL
* International normalized ratio (INR) =< 1.5 (except those subjects who are receiving full-dose warfarin)
* Total bilirubin =< 2.0 mg/dL
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 2.5 times the upper limit of normal for subjects
* Serum creatinine of =< 2.0 mg/dL
* Pregnancy test for women of childbearing potential (serum or urine beta-human chorionic gonadotropin [HCG])
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for four weeks after dosing with AZD6244 ceases; women of child-bearing potential must have a negative pregnancy test prior to entry; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; please note that the AZD6244 manufacturer recommends that adequate contraception for male patients should be used for 16 weeks post-last dose due to sperm life cycle
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD6244 (or its excipient Captisol) or erlotinib
* Previous mitogen-activated protein kinase kinase (MEK) or epidermal growth factor receptor (EGFR) inhibitor use
* Patients with corrected QT (QTc) interval > 480 msecs or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) including heart failure that (i) meets New York Heart Association (NYHA) class III and IV definitions or (ii) is demonstrated by an left ventricular (LV) ejection fraction < 55% on baseline echocardiogram, are excluded
* Required use of a concomitant medication that can prolong the QT interval
* There are potential interactions between erlotinib and cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors and CYP3A4 promoters; although caution and careful monitoring are recommended when use of these compounds is necessary, use of these compounds does not exclude patients from participating in this trial
* Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g. inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; therefore, a negative pregnancy test is required for women of childbearing potential; breastfeeding should be discontinued if the mother is treated with AZD6244
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-11; Primary Completion 2013-04 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ko, Principal Investigator — UCSF-Mount Zion
Locations (2):
- United States (2):
  - UCSF-Mount Zion, San Francisco, California
  - Ohio State University Medical Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Erlotinib Hydrochloride, Selumetinib)
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Erlotinib Hydrochloride, Selumetinib): Patients receive selumetinib by mouth (PO) every day (QD) and erlotinib hydrochloride PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  erlotinib hydrochloride: Given PO
  selumetinib: Given PO
  laboratory biomarker analysis: Correlative studies
Arm/Group | Treatment (Erlotinib Hydrochloride, Selumetinib)
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 67 [40 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 46
Prior chemotherapy [Number; unit: participants]
  Gemcitabine-based | 34
  FOLFIRINOX | 10
  Other | 2
Prior surgery [Number; unit: participants] | 14
Prior radiation [Number; unit: participants] | 7
Elevated baseline Cancer Antigen 19-9(CA19-9) > 2x Upper Limit of Normal (ULN) [Number; unit: participants] | 34
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — Patient Performance Scale:
  0=Fully active, can carry on all pre-disease performance without rest
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair
  5. Dead
  participants
    status = 0 | 32
    status = 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Survival will be calculated according to the method of Kaplan and Meier. Both actual and estimated probability of being alive (along with a 95% confidence interval) at 24 weeks (6 months) and for any multiple of 6 months will be calculated for which the number of uncensored subjects is not smaller than 10.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Erlotinib Hydrochloride, Selumetinib)
Number analyzed (Participants) | 46
months | 7.3 [5.2 to 8.0]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Calculated according to the method of Kaplan and Meier. Actual and estimated probability of being alive and progression-free, along with a 95% confidence interval, will be calculated.
  Response and progression are evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee [JNCI 92(Macdonald et al.):205-216, 2000]. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used. Progressive Disease is defined as a 20% or higher increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: From first dose of study treatment to the date of objective progression, or death due to cancer or unknown cause, or to the date of withdrawal from the trial from unknown reasons, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Erlotinib Hydrochloride, Selumetinib)
Number analyzed (Participants) | 46
months | 1.9 [1.4 to 3.3]

3. Secondary Outcome: CA19-9 Biomarker Response (Defined as a 50% Decline in Serum CA19-9 Level From Baseline in Patients With > 2 x ULN CA19-9 Measurement)
Description: The proportion of patients with CA19-9 response.
Time Frame: Up to 2 years
Population: Patients with baseline levels > 2 x ULN CA19-9 measurement
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Erlotinib Hydrochloride, Selumetinib)
Number analyzed (Participants) | 34
percentage of participants | 38

4. Secondary Outcome: Objective Radiographic Response by RECIST Criteria
Description: Patient's best overall response will be tabulated by level; proportions of complete response (CR) and of CR+partial response will be calculated along with 95% confidence intervals.
  Per Response Evaluation Criteria In Solid Tumors (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR, >= 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR+PR.
Time Frame: Up to 2 years
Population: There were no complete or patial responses by RECIST (stable disease, partial response, or complete response) amongst the 46 participants
Measure: Number; unit: participants
Arm/Group | Treatment (Erlotinib Hydrochloride, Selumetinib)
Number analyzed (Participants) | 46
participants
  Complete Response (CR) | 0
  Complete+Partial Response | 0

5. Secondary Outcome: Incidence of Toxicities Graded Using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: Tabulation of type of adverse events (AE) and the incidence of grade 3 and 4 for each AE
Time Frame: Up to 30 days after completion of study treatment
Measure: Number; unit: events
Arm/Group | Treatment (Erlotinib Hydrochloride, Selumetinib)
Number analyzed (Participants) | 46
events
  Rash | 10
  Diarrhea | 6
  Nausea/vomiting | 4
  Fatigue | 3
  AST/ALT elevation | 4
  Anorexia | 0
  Anemia | 5
  Dysgeusia | 0
  Eye disorders | 0
  Pruritus | 0
  Hypertension | 6
  Thrombocytopenia | 1
  Leukopenia/neutropenia | 1
  Thromboembolic event (incl. cerebral) | 3
  Elevated creatinine | 0

6. Other Pre Specified Outcome: Protein Expression Levels in Pretherapeutic Core Biopsies
Description: Logistic regression models will be used to associate baseline protein markers and best objective response. Cox models will be used to associate baseline protein markers with overall and progression-free survival. Each selected protein markers will be evaluated individually and ranked by the corresponding p-values. Combinations of markers will also be explored.
Time Frame: Up to 2 years
Population: Data was not collected.
Arm/Group | Treatment (Erlotinib Hydrochloride, Selumetinib)
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Circulating Tumor Cell (CTC) Analysis
Description: The association between baseline CTC numbers, their longitudinal changes, and patient outcomes as measured by OS, PFS, and radiographic and biomarker response will be evaluated. The association between expression level of protein markers in CTC with biopsy samples using Pearson's correlation and by unsupervised hierarchical clustering of samples using Pearson correlation as the distance metric will be assessed. Association of longitudinal protein markers in CTC with patient OS will be evaluated using the joint models of longitudinal observations.
Time Frame: Up to 2 years
Population: Data was not collected.
Arm/Group | Treatment (Erlotinib Hydrochloride, Selumetinib)
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Plasma Biomarkers Potentially Predictive of Dual MEK/EGFR Inhibition
Description: The association between candidate plasma biomarkers of interest, their longitudinal changes, and patient outcomes as measured by OS, PFS, and radiographic and biomarker response.
  Specifically, correlation of the relative change in allelic frequency of mutations present in both pre-treatment and on-treatment blood samples versus percent change in CA19-9.
Time Frame: Up to 2 years
Population: Patients who had non-germline mutations (circulating cell-free DNA) represented in both their pre-treatment blood and on-treatment blood samples.
Measure: Number; unit: R^2
Arm/Group | Treatment (Erlotinib Hydrochloride, Selumetinib)
Number analyzed (Participants) | 24
R^2 | 0.1369

9. Primary Outcome: Survival at 24 Weeks
Description: Percent survival at 24 weeks (6 months)
Time Frame: 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Erlotinib Hydrochloride, Selumetinib)
Number analyzed (Participants) | 46
percentage of participants | 58

10. Secondary Outcome: Number of Patients With Dose Modifications and Reason for Dose Modification.
Description: Tabulation of the reasons for dose modification with number of patients
Time Frame: Up to final day of study treatment
Population: Numbers in tabulation total to more than 18 because patients often had 2 or more reasons that prompted dose reduction. For example: Nausea/Vomiting + diarrhea (3), fatigue + diarrhea (2), rash + hypertension (1), rash + diarrhea (1), fatigue + Nausea/Vomiting (1)
Measure: Number; unit: participants
Arm/Group | Treatment (Erlotinib Hydrochloride, Selumetinib)
Number analyzed (Participants) | 18
participants
  RASH | 8
  Diarrhea | 7
  NAUSEA/VOMITING | 5
  Fatigue | 3
  Hypertension | 1
  TRANSAMINITIS | 1
  UNKNOWN | 1

ADVERSE EVENTS:
Arm/Group | Treatment (Erlotinib Hydrochloride, Selumetinib)
Serious Adverse Events (participants affected / at risk) | 22/46
Other Adverse Events (participants affected / at risk) | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Erlotinib Hydrochloride, Selumetinib) (N=46)
Acites (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 4
edema (Blood and lymphatic system disorders) | 1
fatigue (Gastrointestinal disorders) | 11
Platelet count decrease (Blood and lymphatic system disorders) | 1
dehydration (Metabolism and nutrition disorders) | 4
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify - disease progr (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Acute Kidney Injury (Renal and urinary disorders) | 3
Spinal Fracture (Injury, poisoning and procedural complications) | 1
Diarrhea (Gastrointestinal disorders) | 1
Esophageal varicies hemorrhage (Gastrointestinal disorders) | 1
Cardiac disorder (Cardiac disorders) | 1
Pain (General disorders) | 1
anemia (Blood and lymphatic system disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 3
Alanine Aminotransferase increae (Investigations) | 1
Alkaline phosphastase increase (Investigations) | 1
blood bilirubin increase (Investigations) | 1
Aspartate aminotransferase increase (Investigations) | 1
Vaginal infection (Infections and infestations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Chills (General disorders) | 1
Fever (General disorders) | 2
Dypsnea (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal Infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Obstruction gastric (Gastrointestinal disorders) | 1
Confusion - acute dementia (Psychiatric disorders) | 1
Delusion - acute dementia (Psychiatric disorders) | 1
Small intestine ulcer (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Erlotinib Hydrochloride, Selumetinib) (N=46)
Anemia (Blood and lymphatic system disorders) | 13
Elevated white blood cell count (Blood and lymphatic system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Blurred vision (Eye disorders) | 3
Dry eye (Eye disorders) | 1
Left eye irritation (Eye disorders) | 1
Chalazion (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Floaters (Eye disorders) | 2
Photophobia (Eye disorders) | 1
Watering eyes (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 14
Ascites (Gastrointestinal disorders) | 4
Bloating (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 36
Dry Mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 5
Esophageal varices hemorrhage (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal disorders, Other, Specify (Gastrointestinal disorders) | 5
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 25
Obstruction gastric (Gastrointestinal disorders) | 1
Oral dysesthesia (Gastrointestinal disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 1
Small intestine ulcer (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 20
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Chills (General disorders) | 6
Edema face (General disorders) | 1
Edema limbs (General disorders) | 9
Fatigue (General disorders) | 26
Fever (General disorders) | 7
Localized edema (General disorders) | 2
Neck edema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 2
Death NOS (General disorders) | 4
Abdominal infection (Infections and infestations) | 1
Bladder infection (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Paronychia (Infections and infestations) | 3
Skin infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Vaginal infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 2
Spinal fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increase (Investigations) | 13
Alkaline phosphatase increased (Investigations) | 13
Aspartate aminotransferase increased (Investigations) | 21
Blood bilirubin increased (Investigations) | 4
Creatinine increased (Investigations) | 4
INR increased (Investigations) | 3
Investigations - Other, specify (Investigations) | 1
Lymphocyte count decreased (Investigations) | 6
Neutrophil count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 5
Weight loss (Investigations) | 5
White blood cell decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 11
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 11
Tremor (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 2
Delusions (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 4
Hematuria (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Renal and urinary disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 4
Body odor (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 17
Hirsutism (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 10
Rash acneiform (Skin and subcutaneous tissue disorders) | 28
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 15
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 8
Hypotension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
In this single arm, nonrandomized study, an inherent selection bias was likely due to enrollment of patients with favorable disease biology, who had undergone prior resection and fare better compared with those with stage IV disease at diagnosis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less